CLINICAL TRIAL: NCT06324578
Title: A Cross-sectional Observational Study, Based on Immunological and Ultrasonographic Evaluations, to Define the Prevalence of Pre-clinical Sjögren Disease and Other Immune Disturbances in Subjects With Autoimmune Thyroiditis.
Brief Title: Prevalence of Pre-clinical Sjögren Disease and Other Immune Disturbances in Subjects With Autoimmune Thyroiditis Disease
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 25/2023
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-03

CONDITIONS: Sjögren; Autoimmune Thyroid Disease
Keywords: Autoimmune Thyroiditis; Sjögren disease; Immune dysregulation disorders
MeSH Terms: conditions — Sjogren's Syndrome; Thyroiditis, Autoimmune

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- subjects with AT
  Interventions: Diagnostic Test: AT Testing

INTERVENTIONS:
Diagnostic Test: AT Testing — Analysis of blood specimens and neck ultrasonography

SUMMARY:
The main study hypothesis is that Sjögren Disease (SD), usually considered a disorder typical of adult females, may occur not exceptionally in adolescence or even in childhood as a subclinical process. There are several pieces of evidence in favor of this hypothesis, from the incidental detection of asymptomatic SD in pediatric age to biobank-based studies showing that biological signs of SD may precede the disease clinical onset by years or decades. The best scenario to verify this hypothesis could be that of autoimmune thyroiditis, for the following three reasons: 1) subjects with Autoimmune thyroiditis (AT) have a high risk of developing SD (7%); 2) in cases with comorbidity of SD and AT the diagnosis of AT had usually been made before; 3) subjects with AT routinely undergo periodic blood examination and neck ultrasonography (US), which may include Salivary Gland Ultrasound (SGUS) providing contributive data to detect an asymptomatic pre-SD. The knowledge of the real association between AT and pre-SD may impact on several aspects of medicine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 0-17 years with autoimmune thyroiditis
* Subjects between 0-17 years with previous diagnosis of SD or pre-SD

Exclusion Criteria:

* No informed consent from the patient's guardians
* Active or recent infection within one week

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with autoimmune thyroiditis and previous diagnosis of SD or pre-SD
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of pre-SD in pediatric subjects with AT | At the enrolment (T0)
  Pre-SD will be considered in cases with positive Anti-Sjögren's Syndrome A/Anti-Sjögren's Syndrome B antibodies and a positive Outcome Measures in Rheumatology (OMERACT) score at SGUS and/or a "Focus score" ≥1 at labial salivary gland (LSG) or parotid gland biopsy.
  Pre-SD definition meets the American college of rheumatology (ACR)/European league against rheumatism (EULAR) classification criteria for Sjogren Disease if symptoms suspicious of SD are present.
  Non-SD Sialadenitis is defined by a positive SGUS with negative SD related antibodies
Prevalence of pre-SD in pediatric subjects with AT | 12 months after the enrolment (T12)
  Pre-SD will be considered in cases with positive Anti-Sjögren's Syndrome A/Anti-Sjögren's Syndrome B antibodies and a positive Outcome Measures in Rheumatology (OMERACT) score at SGUS and/or a "Focus score" ≥1 at labial salivary gland (LSG) or parotid gland biopsy.
  Pre-SD definition meets the American college of rheumatology (ACR)/European league against rheumatism (EULAR) classification criteria for Sjogren Disease if symptoms suspicious of SD are present.
  Non-SD Sialadenitis is defined by a positive SGUS with negative SD related antibodies
Prevalence of pre-SD in pediatric subjects with AT | 24 months after the enrolment (T24)
  Pre-SD will be considered in cases with positive Anti-Sjögren's Syndrome A/Anti-Sjögren's Syndrome B antibodies and a positive Outcome Measures in Rheumatology (OMERACT) score at SGUS and/or a "Focus score" ≥1 at labial salivary gland (LSG) or parotid gland biopsy.
  Pre-SD definition meets the American college of rheumatology (ACR)/European league against rheumatism (EULAR) classification criteria for Sjogren Disease if symptoms suspicious of SD are present.
  Non-SD Sialadenitis is defined by a positive SGUS with negative SD related antibodies

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste
  - Azienda Sanitaria Universitaria Friuli Centrale (ASU FC), Udine

IPD SHARING:
Plan to Share IPD: Undecided